CLINICAL TRIAL: NCT04766112
Title: Effects of Yang Style Tai Chi Exercises Combined With Mental Imagery Training On Balance and Fall Prevention in Older Adults
Brief Title: Yang Style Tai Chi Exercises Combined With Mental Imagery Training On Balance and Fall Prevention in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00745 Farah Naqvi
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Elderly Population
Keywords: Balance; Yang Style Tai Chi Exercises; mental imagery training; elderly population

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Group I will receive yang style Tai chi exercises combined with mental imagery training which consist of 10 positions
  Interventions: Other: Group II
- Group II (Active Comparator): Group B will receive yang style Tai chi exercise which consist of 10 positions
  Interventions: Other: Group I

INTERVENTIONS:
Other: Group I — Group I will receive yang style Tai chi exercises combined with mental imagery training
  Arms: Group II
Other: Group II — Group II will receive yang style Tai chi exercise which consist of 10 positions.
  Arms: Group I

SUMMARY:
Aging process and the chronic diseases that affect older adults lead to balance disorders, which makes these individuals more susceptible to falls. However, currently there is no evidence available to support effects of Yang Style Tai Chi exercises combined with mental imagery training on balance and fall prevention in older adults. Because separately Tai Chi training techniques having good effects according to evidence .So in this study we will be find out the effects of Tai chi with mental imagery training for the selection of most appropriate treatment method.

DETAILED DESCRIPTION:
Fall is defined as any unintentional positional change that results in a person coming to rest on the ground, floor, or other lower surface. The risk of fall increase dramatically with age. In older adults unintentionally injuries are the fifth leading cause of death, and falls constitute two thirds of these days.

Falls are most serious common condition present in older adults. Falls and balanced problem are more common in elder population, causing injuries, social isolation, and psychological difficulties. Proper balance is imperative for the performance of functional activities. Any deficiency or impairment in balance increases the risk of fall thus making it difficult to perform functional activities. Balance is defined as exertion of postural control that provides a stable base of support while remaining stationary or during movement. Decrease in balance ability resulting from aging triggers motor and gait disabilities in elderly people, which greatly affects their mobility in day-to-day life. They are the serious cause of mortality and morbidity which leads to immobility and premature nursing care.

As life expectancy increases, the problem of falls among the elderly will become more pertinent. Falls occurred in more than one third of the elderly aged 65 years and older annually. The incidence of falls rises steadily from Middle age and peaks in persons older than 80 years. The frequency of falls increases with age and frailty level. Older people who are living in nursing homes fall more often than those who are living in the community. Approximately 30-50% of people living in long term care institutions fall each year, and 40% of them experienced recurrent fall. Approximately 25% to 35% of people over age 65 years experiences more falls every year. Older people have stiffer, less coordinated and more dangerous gaits than younger people. Risk factors for falls among elderly people include environmental hazards and housing characteristic. There are several factors that may influence the fall risk in the elderly to a great extent. Environmental hazards are the leading cause of falls, accounting for about 25 to 45 percent in most studies. Major risk factor of fall among elderly population weakness, mobility impairment, balance and gait disturbance, Dizziness, vertigo, drop attacks, postural hypotension, visual impairment, and syncope are known to cause falls. Attention to these factors significantly reduce the risk of fall. Lower extremity muscle weakness is a significant risk factor for falls, increasing the odds of falling fourfold. A history of fall and gait or balance deficits increases the risk threefold.

Other high-risk situations that can cause or contribute to falls are use of an assistive device, visual deficit, arthritis, and impaired activities of daily living, depression, cognitive impairment, and age older than 80 years. Use of four or more medications has been strongly associated with an increased risk of falls. In particular, use of psychotropic medications, cardiac drugs including class 1A antiarrhythmic agents, digoxin, diuretics, and anticonvulsants have been Implicated in increasing the risk of falls.

There is paucity in the literature regarding evidence for the effectiveness of Tai chi exercises in older adults Lin YC et al 2019 found that in both cross sectional and longitudinal studies that Tai Chi exercises has more effectiveness in balance control, psychological wellbeing ,cardiovascular fitness and postural stability than other exercises. These findings shows that Tai chi exercises has more beneficial and health effective to maintain the good, physical, psychological conditions in older adults.In previous studies have shown beneficial effects of Tai Chi on cardiorespiratory system ,flexibility, Muscle strength, and body fat composition in middle aged and elderly individuals. Likewise, Hong and colleagues found that older adults who had been practicing Tai Chi Chuan for an average of 13.2 years had better balance and functional fitness compared to sedentary older adults. In 2015 Rahal et al in this study 76 elderly individuals who were divided into two groups: the Tai Chi Chuan Group and the Dance Group. The subjects were tested using the Neuro Com Balance MasterH force platform system with the following protocols: static balance testsand dynamic balance tests and found that older expert Tai Chi Chuan practitioners had better bilateral static balance with eyes open on firm and foam surfaces compared to dancers.

A study was done by Cho HY, et al. with the title of Effects of motor imagery training on balance and gait abilities in post-stroke patients published in 2013 and concluded that Adding motor imagery training to gait training produced more significant improvements in the balance and gait abilities than gait training in stroke subjects.

Another study was done by Hamel MF, et al. in 2005 and concluded that the link between attentional demands, postural oscillations, static balance and the prevention of falls among the elderly is of importance. The reduction of attentional demands reflects the automaticity of a task. Therefore, when attentional demands are reduced, more attentional resources are unbound to avoid, among other things, the environmental risk factors that can lead to falls. It has been shown that mental imagery is an effective technique, not only in reducing antero-posterior postural oscillations, but also in interpreting the postural control tasks more automatic. Therefore, this technique may be considered effective among the elderly population, in order to contribute to improving their static balance and preventing falls.

A study was done by Page SJ, et.al with the title of a randomized efficacy and feasibility study of imagery in acute stroke. Published in 2001 and concluded that Imagery technique is a clinically feasible intervention and Imagery, in association with therapy, appears to be a noninvasive, efficacious complement to traditional therapy

ELIGIBILITY:
Inclusion Criteria:

* Age above 60
* Be referred for a fall problem.
* Be identified as being at high risk for a fall on the initial medical assessment (Berg balance scale less than 40/56and at least one accidental fall in the previous 6 month
* Be mentally able to take in an exercise program as assessed with the final SMMSE score is a sum of the 12 items, and can range from a minimum of 0 to a maximum of 30. The SMMSE can be adjusted for non-cognitive disabilities.

Exclusion Criteria:

* Declared unfit for physical activities following medical assessment.
* Present a mental or physical condition incompatible with physical activity.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale: | Change from Baseline , balance to 4Weeks, 8 weeks
  The Berg Balance Scale (BBS) is one of the most widely used tools for balance assessment.
Fall efficacy Scale | Change from Baseline , balance and fall prevention to 4Weeks, 8 weeks
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about falling during 16 social and physical activities inside and outside the home whether or not the person actually does the activity.

SECONDARY OUTCOMES:
Timed Up and Go test (TUG): | Change from Baseline , balance and fall prevention to 4Weeks, 8 weeks
  TUG is a test used to assess a person's mobility. TUG measured the time required for an individual to stand up from a chair with arm rests, walk 3 m, turn, walk back to the chair, and sit down

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Bashart hospital Rawalpindi., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moylan KC, Binder EF. Falls in older adults: risk assessment, management and prevention. Am J Med. 2007 Jun;120(6):493.e1-6. doi: 10.1016/j.amjmed.2006.07.022. PMID 17524747
- [Background] Cameron ID, Dyer SM, Panagoda CE, Murray GR, Hill KD, Cumming RG, Kerse N. Interventions for preventing falls in older people in care facilities and hospitals. Cochrane Database Syst Rev. 2018 Sep 7;9(9):CD005465. doi: 10.1002/14651858.CD005465.pub4. PMID 30191554
- [Background] Ibrahim MS, Mattar AG, Elhafez SM. Efficacy of virtual reality-based balance training versus the Biodex balance system training on the body balance of adults. J Phys Ther Sci. 2016 Jan;28(1):20-6. doi: 10.1589/jpts.28.20. Epub 2016 Jan 30. PMID 26957722
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Voermans NC, Snijders AH, Schoon Y, Bloem BR. Why old people fall (and how to stop them). Pract Neurol. 2007 Jun;7(3):158-71. doi: 10.1136/jnnp.2007.120980. No abstract available. PMID 17515595
- [Background] Blake AJ, Morgan K, Bendall MJ, Dallosso H, Ebrahim SB, Arie TH, Fentem PH, Bassey EJ. Falls by elderly people at home: prevalence and associated factors. Age Ageing. 1988 Nov;17(6):365-72. doi: 10.1093/ageing/17.6.365. PMID 3266440